CLINICAL TRIAL: NCT01230944
Title: Conventional Nissen Fundoplication vs. Laparoscopic Nissen Fundoplication: a Prospective Randomized Study, Long-term Follow-up
Brief Title: Conventional Nissen Fundoplication Versus Laparoscopic Nissen Fundoplication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Paulina Salminen, Turku University Hospital, Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/2004
Record Dates: First submitted 2010-06-24; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: GERD
Keywords: GERD; LNF; CNF; Laparoscopic Nissen fundoplication; Open Nissen fundoplication; Antireflux surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Nissen (Active Comparator): Laparoscopic Nissen fundoplication
  Interventions: Procedure: Laparoscopic Nissen fundoplication
- Open Nissen (Active Comparator): Open (conventional) Nissen fundoplication
  Interventions: Procedure: Open Nissen fundoplication

INTERVENTIONS:
Procedure: Laparoscopic Nissen fundoplication
  Arms: Laparoscopic Nissen
Procedure: Open Nissen fundoplication
  Arms: Open Nissen

SUMMARY:
This is a long-term follow-up of a prospective randomized trial comparing open and laparoscopic Nissen fundoplication.

ELIGIBILITY:
Inclusion Criteria:

* moderate / severe gastrointestinal reflux disease (GERD) requiring operative treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Subjective symptomatic outcome | 15 years
  Evaluation of the symptomatic outcome and the patient satisfaction of the surgical treatment using a structured questionnaire

SECONDARY OUTCOMES:
Endoscopic evaluation of the fundoplication result | 15 years
  Evaluation of the endoscopic objective fudnoplication result by an upper gastrointestinal endoscopy
Reoperation rate | 15 years
Postoperative proton pump inhibitor (PPI) use | 15 years
  postoperative PPI use is registered and the need evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland